CLINICAL TRIAL: NCT01593241
Title: Carboplatin Chemotherapy and Involved Node Radiotherapy in Stage IIA/B Seminoma
Brief Title: Therapy De-escalation in Seminoma Stage IIA/B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Board decided to prematurely terminate the follow-up phase of the trial due to funding reasons
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 01/10; 34569 (Other: SNCTP); 2011-005840-87 (EudraCT Number)
Record Dates: First submitted 2012-05-01; First posted 2012-05-08 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Seminoma
Keywords: Seminoma IIA/B; Carboplatin; RT
MeSH Terms: conditions — Seminoma | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carboplatin (Experimental)
  Interventions: Drug: Carboplatin; Radiation: Involved node RT

INTERVENTIONS:
Drug: Carboplatin — Stage IIA: 1 infusion Carboplatin AUC7 followed by 15 x 2 Gy involved node radiotherapy Stage IIB: 1 infusion Carboplatin AUC7 followed by 18 x 2 Gy involved node radiotherapy
Radiation: Involved node RT — Involved node RT

SUMMARY:
The main objective of this trial is to test the efficacy and safety of carboplatin chemotherapy and involved node radiotherapy in patients with stage IIA/B seminoma.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND

1. Disease background

   Testicular cancers are the most common malignancies in men aged between 18-35 years. Of those, seminoma is the most frequent as it accounts for about half of all testicular cancers. Seminoma is classified according to the involvement of and degree of spreading to lymph nodes and to the lung or other organs. Around 10% of all seminoma patients are diagnosed with stage IIA/B disease. Stage IIA patients have one or more enlarged regional lymph nodes, 2 cm or less in greatest dimension, without evidence of distant disease (cN1 cM0). Stage IIB patients have one or more enlarged regional lymph nodes more than 2 cm but not more than 5 cm in greatest dimension, without evidence of distant disease (cN2 cM0). Paraaortic, interaortocaval, para-/pre-/retrocaval and pre-/retroaortic lymph nodes are considered regional. Intrapelvic, external iliac and inguinal lymph nodes are considered regional only after scrotal or inguinal surgery.

   Seminoma stage IIA/B is highly responsive to chemotherapy or radiation therapy and the progression free survival at 5 or 6 years with such treatments is between 87-95%. Supra-diaphragmatic lymph nodes are the usual site of tumor recurrence after radiation therapy, while local failure or tumor persistence in paraaortic lymph nodes is predominant after chemotherapy.
2. Therapy background

   Current standard of therapy in patients with stage IIA/B seminoma involves either large volume paraaortic and ipsilateral pelvic radiation therapy ("dogleg field") or three cycles of chemotherapy with BEP (Bleomycin, Etoposide, Cisplatin). While both treatment modalities offer high rates of progression free survival and overall survival, they also potentially bear the risk of unwanted events during and following the treatment. Large volume radiation therapy is associated with fatigue, nausea and vomiting during treatment. BEP chemotherapy causes transient fatigue, cytopenia and hair loss. In terms of late adverse events, radiotherapy increases the risk for permanent kidney and bowel damage, while BEP chemotherapy may harm kidneys, lungs, heart and the inner ear. Both therapy modalities may also lead to secondary tumors. Data on late undesirable effects of large field radiation therapy or intensive chemotherapy will become available in the future at the conclusion of long term follow-up analyses of the recent trials. Thus, the current research on seminoma focuses on minimizing short and long term treatment-related morbidity.
3. Previous trials

   Therapy de-escalation has been tested and been proven effective in stage I testicular seminoma patients. For many years, the standard of care for these patients was paraaortic radiation therapy. The trial by Oliver et al. demonstrated the non-inferiority of single dose carboplatin chemotherapy in comparison to paraaortic irradiation in terms of tumor control in patients with stage I seminoma. Although the trial did not present long term data and the demonstration of a lower toxicity profile with carboplatin compared to paraaortic irradiation is still lacking, many clinicians have already switched their treatment strategy to carboplatin chemotherapy in seminoma stage I patients, in hope that this treatment will produce less negative late effects than radiation therapy. Based on these results, we think that a similar therapy de-escalation approach could be attractive in patients with stage II disease.
4. Rationale for performing the trial

Therapy de-escalation for stage IIA/B seminoma has been recently tested in a prospective phase II trial with the use of 3 cycles (for stage IIA) or 4 cycles (for stage IIB) of carboplatin chemotherapy. However, this regime is actually not considered an acceptable treatment because of a relapse rate of 18% at three years. In this trial, all relapsed patients experienced tumor recurrence in the lymph nodes that were initially involved within 3 years following treatment. Thus, while chemotherapy de-escalation with carboplatin leads to a good systemic disease's control, the local control in the involved nodes remains a problem.

On the other hand, no relapse occurs in the initially involved lymph nodes in seminoma IIA/B patients which were treated with large volume irradiation, although 5% of the patients developed distant relapses.

Therefore, one possible way to raise progression free survival in the involved lymph nodes areas to an acceptable level in a therapy de-escalation protocol would be to combine suboptimal carboplatin chemotherapy (1 cycle) with a limited volume of radiation therapy targeting the involved nodes (30 or 36 Gy for stage IIA or IIB, respectively).

It is expected that this combination will trigger less side effects than any of the standard therapies. Previous trials demonstrated that single agent carboplatin is not associated with an increase in the number of adverse events for up to 9 years post chemotherapy. The application of small volume, involved node radiation therapy should avoid damage to viscera and kidneys. Furthermore, the risk for secondary malignancies will likely be reduced because of the low-intensity chemotherapy and dramatically shrunk irradiation field.

This is a single arm trial, in which both stage IIA and IIB patients are included, since all current international treatment recommendations are valid for both disease stages. Selecting exclusively one disease stage for trial inclusion would greatly hamper the feasibility of such a trial.

The trial design, trial treatment and trial specifics are a consensus among the Swiss Urogenital Tumors Project Group, the Swiss Radio-oncology Section and the German Testicular Cancer Study Group.

If the proposed therapy scheme proves to be effective and safe, it will provide a significantly relevant treatment alternative to large volume radiotherapy and intense chemotherapy, and may become the new standard of care for patients with seminoma stage IIA/B.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent before registration.
* Histologically confirmed classical seminoma treated with primary inguinal orchidectomy.
* Tumor stage at diagnosis or at relapse after primary active surveillance is pT1-4* cN1-2 cM0 according to UICC TNM 2009 is pT1-4 cN1-2 cM0 according to UICC TNM 2009.
* Multi-slice CT or MRI or FDG-PET-CT of the chest, abdomen and pelvis or a FDG-PET-CT within 4 weeks prior to patient registration, showing stage IIA/B disease. I.v. contrast medium has to be administered.
* Age ≥ 18 years.
* WHO performance status 0-2.
* Adequate hematological values: neutrophils ≥ 1.0 x 109/L, platelets ≥ 100x 109/L.
* Adequate renal function (calculated creatinine clearance ≥ 50 ml/min, according to the formula of Cockcroft-Gault).
* Patient agrees not to father a child during trial treatment and during 12 months thereafter.
* Patient has been proposed sperm conservation.
* Patient compliance and geographic proximity allow proper staging and follow-up for at least 3 years.

Exclusion Criteria:

* Previous or concurrent malignancy within 5 years with the exception of localized non-melanoma skin cancer or stage I seminoma for patients entering the trial with relapse during active surveillance.
* Psychiatric disorder precluding understanding of information on trial-related topics or giving informed consent or interfering with compliance for treatment schedule.
* Mixed histology seminoma.
* Elevated levels of AFP (≥ULN) at any time.
* Any prior abdominal/pelvic radiotherapy (RT).
* Any anti-cancer therapy after primary tumor resection (active surveillance for stage I disease is not considered as a treatment).
* Any treatment in a clinical trial within 30 days of trial entry.
* Any serious underlying medical condition or serious co-morbidity (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial.
* Any contraindication for the trial drug (for example, known hypersensitivity to trial drug or to any other co-component of the trial drug, past or current renal insufficiency, severe hepatic insufficiency, severe bone marrow dysfunction, tumor bleeding, major hearing defects).
* Any concomitant drugs contraindicated for use with the trial drug according to the approved product information (for example, nephrotoxic or ototoxic medicines).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | at 3 years
  PFS is defined as the time from registration until one of the following events occurs:
  * PD or relapse, defined as progression according to the modified trial-specific version of RECIST 1.1 or a rising level of the tumor marker beta-hCG over the ULN (value must be confirmed by a second measurement). Presence of non-seminoma germ cell tumor has to be excluded in the latter case.
  * Death from any cause.

SECONDARY OUTCOMES:
Adverse events (AEs) temporarily associated with the trial treatment | at 3 years
  AEs are collected from inclusion until 30 days after the end of treatment
Late AEs | at the latest at 20 years
  AEs will be collected from 30 days after the end of treatment until the end of the follow-up phase
Incidence of secondary malignancies | at the latest at 20 years
Response rate | at 3 years
Time to progression (TTP) | at the latest at 20 years
  from registration until documented progressive disease, relapse or death due to tumor.
Overall survival (OS) | at the latest at 20 years.
  from registration to the date of death from any cause
Seminoma specific survival | at the latest at 20 years
  from registration to the date of death due to seminoma
PFS | at the latest at 20 years
  from registration to the date of failure of PFS
Localization of progression | at the latest at 20 years
  from first localization where recurrent tumor disease is detected

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Papachristofilou, MD, Study Chair — University Hospital, Basel, Switzerland; Richard Cathomas, MD, Study Chair — Cantonal Hospital Graubünden; Jens Bedke, Prof, Study Chair — D - University Hospital Tübingen
Locations (25):
- Germany (12):
  - Aachen Universitätsklinik, Aachen
  - Berlin Universitätsklinik Charité, Berlin
  - Berlin Vivantes - Urban, Berlin
  - Berlin Vivantes - Neukölln, Berlin
  - Universitätsklinikum Köln, Cologne
  - Universitaetsklinikum Düsseldorf, Düsseldorf
  - Klinik Essen-Mitte, Essen
  - Hamburg Universitätsklinikum - Eppendorf, Hamburg
  - Krefeld Maria-Hilf Krankenhaus, Krefeld
  - Klinikum Harlaching, München
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Switzerland (13):
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubuenden, Chur
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopital de Sion, Sion
  - Regionalspital Thun, Thun
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papachristofilou A, Bedke J, Hayoz S, Schratzenstaller U, Pless M, Hentrich M, Krege S, Lorch A, Aebersold DM, Putora PM, Berthold DR, Zihler D, Zengerling F, Dieing A, Mueller AC, Schaer C, Biaggi C, Gillessen S, Cathomas R. Single-dose carboplatin followed by involved-node radiotherapy for stage IIA and stage IIB seminoma (SAKK 01/10): a single-arm, multicentre, phase 2 trial. Lancet Oncol. 2022 Nov;23(11):1441-1450. doi: 10.1016/S1470-2045(22)00564-2. Epub 2022 Oct 10. PMID 36228644
- See also: Related Info — http://www.sakk.ch